CLINICAL TRIAL: NCT00321256
Title: Transplantation d'Ilots Pancreatiques Allogeniques Adultes Pour le Traitement du Diabete Insulino-dependant: Etude GRAGIL 2.
Brief Title: Human Islet Transplantation in Brittle Type 1 Diabetes Mellitus. The GRAGIL 2 Study.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Alfediam (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 011226/DGS-2001/0195
Record Dates: First submitted 2006-05-02; First posted 2006-05-03 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: islet transplantation; brittle diabetes; severe hypoglycemia; type 1 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

INTERVENTIONS:
Procedure: human pancreatic islet transplantation

SUMMARY:
This research project is supported by a multicentric network of collaborators whose goal is to assess the efficacy of transplanting allogenic pancreas islets to restore insulin secretion in patients with brittle type 1, insulin-dependent diabetes mellitus and to improve their metabolic control.

DETAILED DESCRIPTION:
The general objective is to demonstrate the beneficial effect of islet allotransplantation in patients with brittle type 1 diabetes with no endogenous insulin secretion, for whom the risk of the spontaneous course of the disease is judged to be worse than the transplantation-related risk. The specific objective is to establish reference data for islet transplantation in non-uremic patients with brittle diabetes, in a multicentric network setting, using the Edmonton protocol.

ELIGIBILITY:
Inclusion criteria:

* Type 1 diabetes mellitus
* Disease duration > 5 years
* Despite intensive insulin therapy with tight endocrinologist supervision, persistence of the following conditions : hypoglycemia unawareness (< 54 mg/dl) ; brittleness with at least two episodes of severe hypoglycemia ((defined by the need for assistance to correct the blood glucose level) or ketoacidosis per year , or often enough that the diabetologist judges the frequency to be life-threatening, the risk of transplantation and immunosuppression being judged to be less than the risk of the spontaneous course of uncontrolled diabetes
* Basal and stimulated plasma C-peptide < 0.2 ng/ml
* Creatinine clearance ≥ 50 ml/min/1.73 m2 and proteinuria < 0.5 g/24h

Exclusion criteria:

* Severe cardiovascular disease (recent myocardial infarction, unstable coronaropathy…)
* Severe systemic infection, including hepatitis C or B viral infection, HIV infection or tuberculosis
* Past or present neoplasia (with the exception of non melanoma skin cancers)
* Body weight > 70 kg in women and BW > 75 kg in men or BMI > 26
* Stimulated C-peptide ≥ 0.3 ng/ml upon Glucagon or Arginine stimulation
* Age < 18 years or > 65 years
* Creatinine clearance < 50 ml/min/1.73 m2
* Albuminuria > 300 mg /24h or proteinuria > 0.5 g/24h
* Hemoglobinemia < 120 g/l in women or < 130 g/l in men
* Liver disease (enzymes > 1.5 N) such as cirrhosis or hepatitis
* Liver hemangioma
* Untreated proliferating diabetic retinopathy
* Pregnancy, lactation, pregnancy project or absence of efficient contraception
* Previous transplantation or immunization as judged by anti-HLA antibodies (> 20%)
* Insulin needs > 0.7 IU/kg/d or > 50 IU
* HbA1c > 12 %
* Any medical condition needing the chronic use of steroids
* Addison disease
* Any hemostasis disorder needing a prolonged treatment with anticoagulation drugs. Low-dose aspirin is permitted. coagulation disorders contraindicating the procedure, such as platelet count < 100000/mm3.
* Serious life-threatening disease
* Medical or surgical history potentially influencing the absorption, distribution, metabolism and clearance of drugs
* Uncontrolled hypercholesterolemia (> 350 mg/dl, 9.1 mmol/l) or hypertriglyceridemia (> 500 mg/dl, 5.6 mmol/l)
* Leukocytes < 4500/mm3, neutrophils < 2000/mm3, platelets < 100000/mm3
* Any medical or psychosocial condition susceptible to interfere with the study, such as drug abuse or recent alcohol abuse
* Poor therapeutic observance
* Failure to communicate or cooperate with the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22
Dates: Start 2003-07; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The rate of insulin-independence, judged upon the following criteria : HbA1c < 6.1%,
post-prandial blood glucose < 180 mg/dl, mean amplitude of glycemic excursion (MAGE index)
< 60 mg/dl, basal C-peptide > 0.5 ng/ml. This insulin independent rate will be assessed 6 months
and 12 months following transplantation.

SECONDARY OUTCOMES:
The rate of success according to the DiaCell composite score defined by the following 4 items : functional islet graft, defined by a basal C-peptide > 0.5 ng/ml;
good metabolic control, defined by HbA1c ≤ 6.5%; disappearance of hypoglycemic events; reduction in exogenous insulin needs ≥ 30%.
Morbidity and quality of life will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Y Benhamou, MD, PhD, Principal Investigator — Universty Hospital, Grenoble, France; Philippe Morel, MD, PhD, Study Chair — University Hospital, Geneva, Switzerland; Charles Thivolet, MD, PhD, Study Director — Hospices Civils de Lyon; Alfred Penfornis, MD, PhD, Study Director — University Hospital, Besancon, France; Laurence Kessler, MD, PhD, Study Director — University Hospital, Strasbourg, France; Eric Renard, MD, PhD, Study Director — University Hospital, Montpellier France; Lionel Badet, MD, PhD, Study Director — Hospices Civils de Lyon; Cyrille Colin, MD, PhD, Study Director — Hospices Civils de Lyon; Thierry Berney, MD, PhD, Study Director — University Hospital, Geneva, Switzerland
Locations (6):
- France (5):
  - University Hospital, Department of Endocrinology, Besançon
  - University Hospital, Department of Endocrinology, Grenoble
  - University Hospital, Department of Endocrinology, Lyon
  - University Hospital, Department of Endocrinology, Montpellier
  - University Hospital, Department of Endocrinology, Strasbourg
- University Hospital, Department of Surgery, Geneva, Switzerland

REFERENCES:
- [Derived] Lablanche S, Borot S, Wojtusciszyn A, Bayle F, Tetaz R, Badet L, Thivolet C, Morelon E, Frimat L, Penfornis A, Kessler L, Brault C, Colin C, Tauveron I, Bosco D, Berney T, Benhamou PY; GRAGIL Network. Five-Year Metabolic, Functional, and Safety Results of Patients With Type 1 Diabetes Transplanted With Allogenic Islets Within the Swiss-French GRAGIL Network. Diabetes Care. 2015 Sep;38(9):1714-22. doi: 10.2337/dc15-0094. Epub 2015 Jun 11. PMID 26068866